CLINICAL TRIAL: NCT02914119
Title: Use of Neuromuscular Blocking Agents and Neuromuscular Monitoring in 7 Danish Teaching Hospitals - a Cross-sectional Study
Brief Title: Use of Neuromuscular Blocking Agents and Neuromuscular Monitoring in 7 Danish Teaching Hospitals
Status: Completed | Type: Observational
Sponsor: Jakob Louis Thomsen (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Jakob Louis Thomsen, MD, Herlev Hospital
Organization: Herlev Hospital (Other)
Other Study IDs: JLT-NM4
Record Dates: First submitted 2016-09-09; First posted 2016-09-26 (Estimated); Results first posted 2019-09-12 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-08

CONDITIONS: Neuromuscular Blockade
Keywords: Residual nerve blockade; Neuromuscular monitoring; Residual curarization; Neuromuscular blocking agents
MeSH Terms: interventions — Rocuronium; Succinylcholine; cisatracurium; Mivacurium; Sugammadex; Neostigmine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Eligible patients: Patients ≥15 years of age who received general anaesthesia with neuromuscular blockade in the last 18 months up until the time of data collection.
  Patients, who are eligible more than once, i.e. undergoing general anaesthesia on more than one occasion, will be included in the analyses as a case for every general anaesthetic received.
  Interventions: Drug: Rocuronium; Drug: Succinylcholine; Drug: Cisatracurium; Drug: Mivacurium; Device: Objective neuromuscular monitoring (acceleromyography); Drug: Sugammadex; Drug: Neostigmine

INTERVENTIONS:
Drug: Rocuronium
Drug: Succinylcholine
Drug: Cisatracurium
Drug: Mivacurium
Device: Objective neuromuscular monitoring (acceleromyography)
Drug: Sugammadex
Drug: Neostigmine

SUMMARY:
Aim: To explore

* the frequency of use of objective neuromuscular monitoring for assessment of depth of neuromuscular blockade in general anaesthesia
* the incidence of residual neuromuscular blockade, and
* the timing of reversal of the neuromuscular blockade at the end of anaesthesia.

We will collect data from 7 Danish anaesthesia departments, using data from the Anaesthesia Information Management System (AIMS).

ELIGIBILITY:
Inclusion Criteria:

Patients who received general anaesthesia with neuromuscular blockade in one of the 7 hospitals providing data for the study in the last 18 months up until the time of data collection

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who received general anaesthesia with neuromuscular blockade
Sampling Method: Non-Probability Sample
Enrollment: 30430 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jakob L Thomsen, MD, Principal Investigator — Sponsor principal investigator
Locations (1):
- Herlev Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No
Sharing of data not included in the permissions granted by authorities stated below

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Estimated number of included cases
Groups:
- Eligible Patients: Patients ≥15 years of age who received general anaesthesia with neuromuscular blockade in the last 18 months up until the time of data collection.
  Patients, who are eligible more than once, i.e. undergoing general anaesthesia on more than one occasion, will be included in the analyses as a case for every general anaesthetic received.
  Rocuronium
  Succinylcholine
  Cisatracurium
  Mivacurium
  Objective neuromuscular monitoring (acceleromyography)
  Sugammadex
  Neostigmine
Period: Overall Study
Arm/Group | Eligible Patients
Started | 30430
Completed | 30430
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Eligible Patients
Number analyzed (Participants) | 30430
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16920
  Male | 13510
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With and Without Objective Neuromuscular Monitoring (Acceleromyography) in Cases Receiving a Non-depolarizing Neuromuscular Blocking Agent (NMBA) (Yes/no)
Time Frame: in the period from induction of anaesthesia to termination of anaesthesia, usually 2 hours
Population: Patients receiving non-depolarizing neuromuscular blocking agent
Measure: Count of Participants; unit: Participants
Arm/Group | Eligible Patients
Number analyzed (Participants) | 16525
Participants
  Monitoring applied | 14463
  Monitoring not applied | 2062

2. Primary Outcome: Number of Participants With and Without Objective Neuromuscular Monitoring (Acceleromyography) in Cases Receiving a Depolarizing NMBA (Succinylcholine) (Yes/no)
Time Frame: in the period from induction of anaesthesia to termination of anaesthesia, usually 2 hours
Population: Patients receiving succinylcholine only
Measure: Count of Participants; unit: Participants
Arm/Group | Eligible Patients
Number analyzed (Participants) | 13905
Participants
  Monitoring applied | 4224
  Monitoring not applied | 9681

3. Secondary Outcome: Last Recorded Train-of-four (TOF) Ratio Before Tracheal Extubation or Removal of Supraglottic Airway Device in Patients Receiving a Non-depolarizing NMBA
Description: The train-of-four (TOF) ratio is the ratio between the last and first measurements after four stimuli of the ulnar nerve at 2 Hz. The ratio should be at least 0.9 before tracheal extubation.
Time Frame: in the period from induction of anaesthesia to termination of anaesthesia, usually 2 hours
Population: Only participants with data on the outcome was analyzed, as per protocol.
Measure: Median (Inter-Quartile Range); unit: Train-of-four ratio
Arm/Group | Eligible Patients
Number analyzed (Participants) | 16525
Train-of-four ratio | 0.97 [0.90 to 1.06]

4. Secondary Outcome: Number of Participants With and Without Administration of Sugammadex in Cases Receiving a Non-depolarizing NMBA (Yes/no)
Time Frame: in the period from induction of anaesthesia to discharge from the post-anaesthesia care unit, usually 5 hours
Population: Only participants with data on the outcome was analyzed, as per protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Eligible Patients
Number analyzed (Participants) | 13090
Participants
  Yes | 145
  No | 12945

5. Secondary Outcome: Number of Participants With and Without Administration of Neostigmine in Cases Receiving a Non-depolarizing NMBA (Yes/no)
Time Frame: in the period from induction of anaesthesia to discharge from the post-anaesthesia care unit, usually 5 hours
Population: Only participants with data on the outcome was analyzed, as per protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Eligible Patients
Number analyzed (Participants) | 16525
Participants
  Yes | 8570
  No | 7955

6. Secondary Outcome: Time in Minutes From Tracheal Extubation or Removal of Supraglottic Airway Device to Discharge From Post-anaesthesia Care Unit in Cases Involving a Non-depolarizing NMBA With and Without Neuromuscular Monitoring, Respectively
Time Frame: in the period from induction of anaesthesia to discharge from the post-anaesthesia care unit, usually 180 minutes
Population: Only participants with data on the outcome was analyzed, as per protocol.
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Eligible Patients
Number analyzed (Participants) | 12700
Minutes | 97 [63 to 157]

7. Secondary Outcome: Number of Participants With and Without Mild Oxygen Desaturation (<90%, But >80%) in Cases Receiving a Non-depolarizing NMBA
Time Frame: in the period between tracheal extubation or removal of supraglottic airway device and discharge from post-anaesthesia care unit, assessed up to 24 hours
Population: Only participants with data on the outcome was analyzed, as per protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Eligible Patients
Number analyzed (Participants) | 15983
Participants
  Desaturation | 1753
  No desaturation | 14230

8. Secondary Outcome: Number of Participants With and Without Severe Oxygen Desaturation (<80%) in Cases Receiving a Non-depolarizing NMBA
Time Frame: as for outcome 7
Population: Only participants with data on the outcome was analyzed, as per protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Eligible Patients
Number analyzed (Participants) | 15983
Participants
  Desaturation | 295
  No desaturation | 15688

ADVERSE EVENTS:
Time Frame: Averse events data were not collected for the study because it was a retrospective database study. Adverse events were collected and reported by individual institutions according to local procedure.
Description: Averse events data were not collected for the study because it was a retrospective database study. Adverse events were collected and reported by individual institutions according to local procedure.
Arm/Group | Eligible Patients
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-08-03): https://cdn.clinicaltrials.gov/large-docs/19/NCT02914119/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-03): https://cdn.clinicaltrials.gov/large-docs/19/NCT02914119/SAP_001.pdf